CLINICAL TRIAL: NCT00001836
Title: Detection of Coronary Artery Calcification: Comparison of Volumetric and Electron Beam Computed Tomography
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990001; 99-CC-0001
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-11

CONDITIONS: Coronary Disease
Keywords: Coronary Artery Disease; EBCT; Volumetric Scan; Coronary Artery Calcium; Prospective Gating
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

SUMMARY:
Electron beam computed tomography (EBCT) has been regarded as the state-of-the-art investigation for detecting and quantitating coronary artery calcification. However, EBCT is expensive, and the asymmetric gantry geometry makes it less useful for routine scanning; thus, EBCT is not readily available to the general population. Recent reports have shown that "volumetric" (also known as "helical" or "spiral") scanners, which are much more commonly available than EBCT, can detect coronary artery calcifications. Updated software available to the NIH which will allow for EKG gating of volumetric scans should improve the quality of the images, and thus improve the ability to accurately quantitate coronary calcification by volumetric scanners. We would like to compare the results of volumetric scans with that of standard EBCT in order to characterize similarities and differences between the two scanning techniques. We propose to obtain EBCT and volumetric CT scans of the coronary arteries in a group of patients with known or suspected coronary artery disease and to calculate the calcium score by each method. Our primary analysis will be a comparison of the sensitivities of the two methods.

DETAILED DESCRIPTION:
Electron beam computed tomography (EBCT) has been regarded as the state-of-the-art investigation for detecting and quantitating coronary artery calcification. However, EBCT is expensive, and the asymmetric gantry geometry makes it less useful for routine scanning; thus, EBCT is not readily available to the general population. Recent reports have shown that "volumetric" (also known as "helical" or "spiral") scanners, which are much more commonly available than EBCT, can detect coronary artery calcifications. Updated software available to the NIH which will allow for EKG gating of volumetric scans should improve the quality of the images, and thus improve the ability to accurately quantitate coronary calcification by volumetric scanners. We would like to compare the results of volumetric scans with that of standard EBCT in order to characterize similarities and differences between the two scanning techniques. We propose to obtain EBCT and volumetric CT scans of the coronary arteries in a group of patients with known or suspected coronary artery calcification, including subjects of sufficiently advanced age, and to calculate the calcium score by each method. Our primary analysis will be a comparison of the sensitivities of the two methods.

ELIGIBILITY:
Must have known or suspected coronary artery calcification, including subjects of age equal to or greater than 55 years (men), or 65 years (women).

Must be at increased risk for CAD. (Chronic hypertension greater than 140/90, cholesterolemia greater than 130 mg/dl, active cigarette smoker, or diabetes mellitus.)

Must be 18 years of age or older.

Females must not be pregnant or considering pregnancy and must not be lactating.

Must not have any surgical devices which may interfere with imaging: heart valves, pacemakers, sternal wire sutures, epicardial pacer leads, metallic coronary stents.

Must not have tachycardia greater than 90 bpm at time of scanning, or other fast or irregular rhythm.

Must not be obese. Patients weighing more than 300 pounds will be excluded since this is the table weight limit for the EBCT scanner.

Must be able to suspend respiration for 28 seconds at time of scanning.

Must be able to give informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 213
Dates: Start 1998-10; Study Completion 2001-11

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Breen JF, Sheedy PF 2nd, Schwartz RS, Stanson AW, Kaufmann RB, Moll PP, Rumberger JA. Coronary artery calcification detected with ultrafast CT as an indication of coronary artery disease. Radiology. 1992 Nov;185(2):435-9. doi: 10.1148/radiology.185.2.1410350.
- [Background] Kaufmann RB, Sheedy PF 2nd, Breen JF, Kelzenberg JR, Kruger BL, Schwartz RS, Moll PP. Detection of heart calcification with electron beam CT: interobserver and intraobserver reliability for scoring quantification. Radiology. 1994 Feb;190(2):347-52. doi: 10.1148/radiology.190.2.8284380.
- [Background] Shemesh J, Apter S, Rozenman J, Lusky A, Rath S, Itzchak Y, Motro M. Calcification of coronary arteries: detection and quantification with double-helix CT. Radiology. 1995 Dec;197(3):779-83. doi: 10.1148/radiology.197.3.7480756.